CLINICAL TRIAL: NCT04389060
Title: Effects of Acute Grape Seed Extract Supplementation on Hemodynamics in Obese Males
Brief Title: Effect of Acute Dietary Supplementation With Grape Seed Extract on Aortic Stiffness, Arterial Pressure, and Blood Vessel Dilation in Collegiate Obese Individuals at Rest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Principal Investigator, Jong-Kyung Kim, Associate Professor, California Baptist University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 081-1819-EXP
Record Dates: First submitted 2020-05-08; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind, cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSE group (Active Comparator): Subjects took a single dose of 600 mg GSE in capsule form through ingestion 2 hours prior to testing
  Interventions: Dietary Supplement: Grape seed extract
- Placebo group (Placebo Comparator): Subjects took a single dose of 600 mg starch in capsule form through ingestion 2 hours prior to testing
  Interventions: Dietary Supplement: Grape seed extract

INTERVENTIONS:
Dietary Supplement: Grape seed extract — Two capsule grape seed extract (total 600 mg)

SUMMARY:
This study investigated if elevated BP and aortic stiffness characterized in obese individuals are attenuated following acute grape seed extract supplementation. It is hypothesized that acute dietary supplementation with grape seed extract attenuates aortic stiffness, systolic blood pressure, diastolic blood pressure, mean arterial pressure, and total peripheral resistance and these effects are partially due to reductions in peripheral vasoconstriction

DETAILED DESCRIPTION:
Twenty men (obese = 10; normal body weight (NBW) = 10) participated in this study. Effects of placebo (PL: 600 mg) and GSE (600 mg) on systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (Q), total peripheral resistance (TPR), and AoS were compared 2 h after ingestion of GSE or PL on different days, one week apart. Arterial blood pressure was measured using a sphygmomanometer from a brachial artery at the level of the heart on chair. HR and SV were continuously measured using a non-invasive device (Physio Flow). CO was calculated by HR X SV. TPR was calculated by MAP/CO.

ELIGIBILITY:
Inclusion Criteria:

* Obesity: body mass index (>30), Normal body weight: body mass index (25-29)

Exclusion Criteria:

* cardiovascular diseases or consume any antihypertensive medication or supplementation that can affect blood pressure or aortic stiffness

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
change in heart rate | 2 hours after each supplementation
  beats per minute
change in stroke volume | 2 hours after each supplementation
  volume per stroke
change in cardiac output | 2 hours after each supplementation
  total volume for a minute
change in systolic blood pressure | 2 hours after each supplementation
  pressure exerted during contraction
change in diastolic blood pressure | 2 hours after each supplementation
  pressure exerted during relaxation
change in mean arterial pressure | 2 hours after each supplementation
  One reported pressure (systolic blood pressure-diastolic blood pressure)/3 + diastolic blood pressure
change in total peripheral resistance | 2 hours after each supplementation
  One reported value (mean arterial pressure/cardiac output)

CONTACTS AND LOCATIONS:
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided